CLINICAL TRIAL: NCT05051202
Title: A Randomised, Single-blind, Comparator-controlled, Crossover Study, Assessing the Tolerable Upper Intake Level and Safety of Sugars From Fiber in Healthy Adults
Brief Title: A Study Assessing the Tolerable Upper Intake Level and Safety of Sugars From Fiber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Glycoscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CG1141
Record Dates: First submitted 2021-06-14; First posted 2021-09-21 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Gastrointestinal Tolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 25g Sugars From Fiber per day (Experimental): Administered in 50 g Flapjacks containing 25 g Fiber (from Sugars from Fiber), taken 3 times per day, after meals, for a 14 day period
  Interventions: Other: Sugars from Fiber
- 25g Resistant Maltodextrin per day (Active Comparator): Administered in 50 g Flapjacks containing 25 g Resistant Maltodextrin, taken 3 times per day, after meals, for a 14 day period
  Interventions: Other: Resistant Maltodextrin
- 35g Sugars From Fiber per day (Experimental): Administered in 50 g Flapjack containing 35 g Fiber (from Sugars from Fiber), taken 3 times per day, after meals, for a 14 day period
  Interventions: Other: Sugars from Fiber
- 35g Resistant Maltodextrin per day (Active Comparator): Administered in 50 g Flapjacks containing 35 g Resistant Maltodextrin, taken 3 times per day, after meals, for a 14 day period
  Interventions: Other: Resistant Maltodextrin
- 45g Sugars From Fiber per day (Experimental): Administered in 50 g Flapjacks containing 45 g Fiber (from Sugars from Fiber), taken 3 times per day, after meals, for a 14 day period
  Interventions: Other: Sugars from Fiber
- 45g Resistant Maltodextrin per day (Active Comparator): Administered in 50 g Flapjacks containing 45 g Resistant Maltodextrin, taken 3 times per day, after meals, for a 14 day period
  Interventions: Other: Resistant Maltodextrin

INTERVENTIONS:
Other: Sugars from Fiber — Proprietary blend of Sugars from Fiber baked into 50 g flapjack
  Other Names: SFF
  Arms: 25g Sugars From Fiber per day; 35g Sugars From Fiber per day; 45g Sugars From Fiber per day
Other: Resistant Maltodextrin — Resistant Maltodextrin baked into 50 g flapjack
  Other Names: RM
  Arms: 25g Resistant Maltodextrin per day; 35g Resistant Maltodextrin per day; 45g Resistant Maltodextrin per day

SUMMARY:
The purpose of this study is to determine the upper tolerable limit of Sugars from Fiber

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent;
* Be between 18 and 60 years of age inclusive;
* Have a body mass index <30 Kg/m2;
* Be in general good health, as determined by the investigator;
* Have a habitual dietary intake of ≥13g fibre/day;
* Self-reported consumption of a generally 'healthy diet'.

Exclusion Criteria:

* Females who are pregnant, lactating or wish to become pregnant during the study;
* Participant has self-reported low-energy diet or other extreme dietary habits;
* Have experienced recurrent loose stool within the past 4 weeks;
* Recent gastroenteritis or food borne illness such as confirmed food poisoning within the past 4 weeks;
* Have taken a medication or dietary supplement that may influence GI activity within the 2-weeks prior to screening;
* Have a history of abdominal surgery (excluding appendectomy);
* Have taken anaesthesia within the past 4 weeks;
* Have a known or suspected food allergy or intolerance to any of the investigational product ingredients;
* Have taken antibiotics within the past 12-weeks;
* Have a recent history of drug and/or alcohol abuse at the time of enrolment;
* Are a smoker (defined as >5 cigarettes/week);
* Have made any major dietary change in the past 3 months;
* Have planned major changes in lifestyle (i.e. diet, dieting, exercise level, travelling) during the duration of the study;
* Have an active gastrointestinal disorder or previous gastrointestinal surgery;
* Have irritable bowel syndrome, diagnosed or undiagnosed and treated with chronic medications;
* Have a gastrointestinal disease i.e., chronic diarrhoea, Crohn's disease, ulcerative colitis, diverticulosis, stomach or duodenal ulcers, or with a history of such diseases;
* Have a metabolic or endocrine disorder such as diabetes, thyroidism, or other metabolic disorder;
* Have a severe chronic disease i.e. cancer, renal failure, hepatitis, HIV, cirrhosis etc., or with a history of such diseases;
* Are severely immunocompromised (HIV positive, transplant patient, on antirejection medications, on a systemic steroid for >30 days, or chemotherapy or radiotherapy within the last year);
* Have a personal history of anorexia nervosa, bulimia, or significant eating disorders;
* Experiences alarm features such as unintentional weight loss, rectal bleeding, recent change in bowel habit (<3 months) or abdominal pain;
* Participants who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial;
* Participant is currently receiving treatment involving experimental drugs. If the participant has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in the composite score of gastrointestinal symptoms, (bloating score + abdominal cramping score + stomach noises score + flatulence score), in the treatment groups as compared to control, reported daily in the eDiary | 14 days
  Participants rate each symptom on a 0-5 scale (0 = no symptoms; 5 = severe symptoms). A sum of each of the symptom scores is calculated minimum possible score is 0 and maximum is 30. Higher scores indicate worsening Gastrointestinal symptoms.

SECONDARY OUTCOMES:
Incidence of Type 6 (Fluffy pieces with ragged edges - a mushy stool) or Type 7 (Watery, no solid pieces - entirely liquid) Bristol Stool Scale score, in the treatment groups as compared to control, recorded daily in the eDiary. | 14 days
  Participants will identify each bowel movement 'type' using the Bristol Stool Scale (Type 1 = hard stool difficult to pass [classified as severe constipation]; Type 7 = watery, entirely liquid stool [classified as severe diarrhea]). 'Normal' stool is considered to be Types 3 and 4; Type 5 would suggest the participant lacks dietary fiber, and Types 6 and 7 would be considered to suggest mild and severe diarrhea, respectively. This endpoint will show the incidence of participants experiencing 'diarrhea' Type stool. A lower incidence of diarrhea-type stools would indicate higher fiber content in the groups diet.
Difference in mean and highest Bristol Stool Scale score, in the treatment groups as compared to control, reported daily in the eDiary | 14 days
  Participants will identify each bowel movement 'type' using the Bristol Stool Scale (Type 1 = hard stool difficult to pass [classified as severe constipation]; Type 7 = watery, entirely liquid stool [classified as severe diarrhea]). 'Normal' stool is considered to be Types 3 and 4; Type 5 would suggest the participant lacks dietary fiber, and Types 6 and 7 would be considered to suggest mild and severe diarrhea, respectively. Lower 'types' are indicative of constipation, and higher 'types' are indicative of diarrhea.
Difference in mean stool frequency, in the treatment groups as compared to control, reported daily in the eDiary | 14 days
  Participants will identify each bowel movement 'type' using the Bristol Stool Scale (Type 1 = hard stool difficult to pass [classified as severe constipation]; Type 7 = watery, entirely liquid stool [classified as severe diarrhea]). 'Normal' stool is considered to be Types 3 and 4; Type 5 would suggest the participant lacks dietary fiber, and Types 6 and 7 would be considered to suggest mild and severe diarrhea, respectively. Lower 'types' are indicative of constipation, and higher 'types' are indicative of diarrhea.
Absolute change in Gastrointestinal Symptom Rating Scale (GSRS) total score, in the treatment groups as compared to control, from baseline to Day 7 of intervention | 14 days
  The Gastrointestinal Symptom Rating Scale questionnaire contains 15 items, each uses a seven-graded Likert scale, where 1 represents the most positive option (no symptoms) and 7 the most negative one (severe symptoms). The participant will answer each question with respect to their experience over the last 7 days. To calculate the Total Score, each of the 15 item scores will be used to calculate a mean Total Score: minimum possible score = 0; maximum possible score = 7; higher scores indicate worse symptoms.
  As the recall period is 7 days, the Baseline value will give a score from Day -6 to Day 0, and the Day 7 value will give a score from Day 1 to Day 7 - a 14 day period overall.
Absolute change in GSRS total score, in the treatment groups as compared to control, from baseline to Day 14 of intervention | 14 days
  The Gastrointestinal Symptom Rating Scale questionnaire contains 15 items, each uses a seven-graded Likert scale, where 1 represents the most positive option (no symptoms) and 7 the most negative one (severe symptoms). The participant will answer each question with respect to their experience over the last 7 days. To calculate the Total Score, each of the 15 item scores will be used to calculate a mean Total Score: minimum possible score = 0; maximum possible score = 7; higher scores indicate worse symptoms.
  As the recall period is 7 days, the Baseline value will give a score from Day -6 to Day 0, and the Day 7 value will give a score from Day 1 to Day 7 - a 14 day period overall.
Percentage of Participants with worsening GSRS scores between Baseline (Day 0) and Day 14 compared to between Day 21 and Day 35 in the treatments group as compared to control | 14 days
  The Gastrointestinal Symptom Rating Scale questionnaire contains 15 items, each uses a seven-graded Likert scale, where 1 represents the most positive option (no symptoms) and 7 the most negative one (severe symptoms). The participant will answer each question with respect to their experience over the last 7 days. To calculate the Total Score, each of the 15 item scores will be used to calculate a mean Total Score: minimum possible score = 0; maximum possible score = 7; higher scores indicate worse symptoms.
  As the recall period is 7 days, the Baseline value will give a score from Day -6 to Day 0, and the Day 7 value will give a score from Day 1 to Day 7 - a 14 day period overall.
Difference in severity and frequency of related AEs in the treatment groups as compared to control, reported in the AE Log | 14 days
Incidence of out of range blood safety parameters (Chemistry and FBC), in the treatment groups as compared to control, from baseline to Day 14 of intervention | 14 days
  This outcome will report the incidence of 'out of range' blood safety parameters assessed from a standard safety chemistry panel (ALT, AST, BUN, Chloride, Creatinine, Potassium, Protein, Sodium) and a standard safety hematology panel (WBC, RBC, Hemoglobin, Hematocrit, Platelets, MCV, MCH, MCHC, RDW). 'Out of range' is determined based on clinically defined 'normal' ranges for each analyte. A higher incidence of 'out of range' blood safety parameters would be a worse safety outcome in this case.
Incidence of out of range Urinalysis safety parameters in the treatment groups as compared to control, from baseline to Day 14 of intervention | 14 days
  This outcome will report the incidence of 'out of range' Urinalysis safety parameters (Glucose, Bilirubin, Ketone, Specific Gravity, Blood, pH, Protein, Urobilinogen, Nitrite and Leukocyte Esterase). 'Out of range' is determined based on clinically defined 'normal' ranges for each analyte. A higher incidence of 'out of range' urinalysis safety parameters would be a worse safety outcome in this case.
Absolute change in systolic blood pressure (mmHg) in the treatment groups as compared with control, from baseline to Day 14 of intervention | 14 days
Absolute change in diastolic blood pressure (mmHg) in the treatment groups as compared with control, from baseline to Day 14 of intervention | 14 days
Absolute change in heart rate (BPM) in the treatment groups as compared with control, from baseline to Day 14 of intervention | 14 days
Absolute change in body temperature (˚C) in the treatment groups as compared with control, from baseline to Day 14 of intervention | 14 days

OTHER OUTCOMES:
Change in fecal Short Chain Fatty Acids (fSCFA) microbiota, in the treatment groups as compared with control, from baseline to Day 14 of intervention | 14 days
Change in Faecal pH, in the treatment groups as compared with control, from baseline to Day 14 of intervention | 14 days
Change in microbial community analysed using Shallow Shotgun Sequencing, in the treatment groups as compared with control, from baseline to Day 14 on intervention | 14 days
Detection of oligosaccharides in plasma at Day 14 on intervention. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, Ph.D, Principal Investigator — Atlantia Food Clinical Trials
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moura de Oliveira Beltrame D, Simmons TJ, Jenkins AL, Dinan T, Nicholson TJ. Gastrointestinal Tolerability and Acute Glycemic Response of Oligosaccharides and Polysaccharides from Cellulose and Xylan in Healthy Adults: Two Double-Blinded, Randomized, Controlled, Cross-over Trials. J Am Nutr Assoc. 2024 May-Jun;43(4):305-314. doi: 10.1080/27697061.2023.2282615. Epub 2023 Nov 30. PMID 38032277